CLINICAL TRIAL: NCT04779372
Title: Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) for Chronic Insomnia ：A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Zeen health (Beijing) Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Jing MA, Dr., Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-773
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Insomnia
Keywords: Insomia, CBTI, Online treatment, Telemedicine, Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be random allocation into two groups named Group dCBT-I and Group Sleep Education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of dCBT-I (Experimental): participants will receive 6-week smartphone-based dCBT-I from a Wechat applet
  Interventions: Behavioral: smartphone-based dCBT-I from a Wechat applet
- Group of sleep education (Sham Comparator): Patients will receive sleep health education like the advices getting from common sleep clinic by the same applet as the group of CBT-I in smartphone
  Interventions: Behavioral: sleep education

INTERVENTIONS:
Behavioral: smartphone-based dCBT-I from a Wechat applet — Participants will receive 6-week smartphone-based dCBT-I from a Wechat applet.
  Arms: Group of dCBT-I
Behavioral: sleep education — Participants will receive sleep education like the advices getting from common sleep clinic.
  Arms: Group of sleep education

SUMMARY:
This randomized, open, parallel controlled study aims to explore the clinical effectiveness of smartphone-based digital Cognitive behavioural therapy for insomnia（dCBT-I）. Patients who diagnosed chronic insomnia disorder and proficient in using mobile phone intended to receive CBT-I. Participants will be random allocation into Group dCBT-I and Group Sleep Education. Primary outcome is the insomnia severity as measured using the Insomnia Severity Index (ISI).

DETAILED DESCRIPTION:
This is a single-center, randomized, open, parallel controlled study. Patients who had no CBTI treatment before for chronic insomnia will be recruited and followed for 6 weeks. Participants will be random allocation into Group dCBT-I and Group Sleep Education, and then explore the clinical effectiveness of smartphone-based digital CBT-I therapy. We will collect the baseline information: population characteristics, including age, sex, education, employment, living and residential status, demographic data, smoking and alcohol consumption, body mass index (BMI); medical history and medication status and adverse reactions during treatment. Primary outcome is the Insomnia Severity Index (ISI). Secondary outcomes include an online sleep diary measured information regarding: time in bed(TIB), total sleep time (TST), sleep efficiency (SE), total wake time(TWT); bracelet measured information regarding: total sleep time (TST), sleep latency(SL), sleep efficiency (SE), the times of wake from sleep(TWS), sleep quality score setting by bracelet; the 16-item Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16); Fatigue Severity Scale(FSS); Health-related Quality of Life (SF-12); Generalized Anxiety Disorder Scale-7 (GAD-7); Patient Health Questionnaire-9 (PHQ-9).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18y;
2. Participants who meet proposed ICSD-3 and DSM-5 criterias for persistent Insomnia Disorder. (a) a current complaint of poor sleep (diffculty initiating and/or maintaining sleep, early morning wakening, or non-restorative sleep); with (b) signifcant daytime effects in 1 of 6 domains (fatigue, daytime sleepiness, cognitive impairment [e.g., concentration problems], mood disturbance, impaired occupational or academic functioning [e.g., poor productivity], impaired interpersonal/ social functioning); and (c) affecting them 3 nights per week for 3 months.
3. Insomnia Severity Index (ISI) ≥14;
4. If a comorbid sleep or psychiatric disorder is present, treatment of this condition should be stable at the time of entry in the study. There is no requirement of insomnia medications.
5. Can use APP/ Wechat applet skillfully, can freely communicate, read and fill the electronic questionnaire, well understanding.
6. Sign informed consent

Exclusion Criteria:

1. The presence of shift work, head injury, acute suicidality, current mania, schizophrenia or elevated substance use.
2. With documented severe physical diseases impairing sleep: such as craniocerebral disease, cancer pain, unstable angina or uncontrolled heart failure, etc.
3. Current or past CBT-I
4. Epworth Sleepiness Scale (ESS) ≥12
5. Without informed consent or not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | V2 and V4 visit ( 6, 18 weeks after recruitment).
  The ISI is a 6-item self-report measure of impairment in daytime functioning due to inadequate sleep. The ISI shows adequate internal consistency, appropriate test-retest reliability, and sensitivity to change with treatment. Scores can range from 0 to 28, with higher scores indicating more impairment. Scores higher than 14 are thought to be indicative of the presence of clinical insomnia and change in scores of 8.4 have been found to reflect moderate improvement in clinical samples.

SECONDARY OUTCOMES:
Sleep characters recorded by online sleep diary | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  Participants will be encouraged to record sleep diaries each day duration the 6-week of intervention. Participants will complete 7-day online sleep diaries at baseline before recruitment, and 1month, 3month and 6month after intervention. The following parameters extracted from the diary will be used for analysis: time in bed(TIB), total sleep time (TST), sleep latency(SL), sleep efficiency (SE), the times of wake from sleep(TWS), self-scored sleep quality. Data suggest that tracking sleep parameters through these diaries can provide a more comprehensive understanding of sleep status.
Sleep characters recorded by smart bracelet | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  The participants will wear the bracelet everyday at each evaluating time point for at least week before each evaluation/visit. The following parameters recorded by the bracelet will be used for analysis: total sleep time (TST), sleep latency(SL), sleep efficiency (SE), the times of wake from sleep(TWS), sleep quality score setting by bracelet.
Dysfunctional Beliefs and Attitudes about sleep scale (DBAS-16) | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  All items in DBAS-16 will be answered on a 10-point Likert scale ranging from 0 (strongly disagree) to 10 (strongly agree). As emphasized by Morin et al, there is no absolute right or wrong answer for a single item. Rather, the degree to which a particular item is endorsed by a participant is a reflection of the nature of the dysfunction. The mean scores are summed to generate a DBAS-16 overall index and four subscales (consequences, worry/helplessness, expectations, medication), with higher scores reflecting stronger dysfunctional beliefs and attitudes about sleep.
Fatigue Severity Scale(FSS) | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  The scale employs nine items to measure the self-reported impact of fatigue. Responses to individual items are rated on a 7-point Likert scale, ranging from 1 = strongly disagree to 7 = strongly agree. The FSS score is calculated as the mean of all item scores, with a score of C4 indicating abnormal fatigue and a score of C5 indicating severe fatigue.
Health-related Quality of Life (SF-12) | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  The SF-12 derived from the SF-36 and measured Quality of Life with 12 items. It generates a profile of respondents HRQoL across eight domains: physical function (PH), role physical (RP), bodily pain (BP), general health (GH), vitality (V), social function (SF), role emotion (RE), and mental health (MH). Finally, the SF-12 generates a summary of physical functional scores (PCS) and mental functional scores (MCS). The PCS is calculated based on a combination of physical functioning, role physical, bodily pain and general health scores. The MCS is calculated based on a combination of vitality, social functioning, role emotional, and mental health scores.
Generalized Anxiety Disorder Scale-7 (GAD-7) | baseline, and 6, 10,18, 30 weeks after recruitment. Some participants 52 weeks after recruitment decided by themselves.
  The GAD-7 is designed for use in primary care patients. The GAD-7 consists of a self-report questionnaire that allows for the rapid detection of GAD. Subjects will be asked if they are bothered by anxiety related problems over the past two weeks by answering seven items on a 4-point scale. The total scores range from 0 to 21. At a cutoff score of 9, the GAD-7 has a sensitivity of 89 % and a specificity of 82 % for detecting GAD compared with a structured psychiatric interview.
Insomnia Severity Index (ISI) at V3 and V5 visit | V3 and V5 visit ( 10, 30 weeks after recruitment).
  The comparisons of ISI between CBT-I and control group at V3 and V5 visit
Insomnia Severity Index (ISI) improvement | 6, 10,18, 30 weeks after recruitment.
  Comparisons of ISI improvement values, improvement rate, treatment response rate and insomnia remission rate between dCBT-I group and control group
Patient Health Questionnaire-9 (PHQ-9) | baseline, and 6, 10,18, 30 weeks after recruitment.
  The PHQ-9 is a self-report measure of depression used widely in research and as a screening measure in primary care and hospital settings.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Doctor, Study Chair — Peking University First Hospital; Cheng Zhang, Doctor, Study Director — Peking University First Hospital; Yanan Liu, Doctor, Study Director — Peking University First Hospital; Yane Shen, Postgraduate, Study Director — Peking University First Hospital; Xiaoming Guo, Doctor, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang C, Liu Y, Guo X, Liu Y, Shen Y, Ma J. Digital Cognitive Behavioral Therapy for Insomnia Using a Smartphone Application in China: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e234866. doi: 10.1001/jamanetworkopen.2023.4866. PMID 36972049